CLINICAL TRIAL: NCT03971994
Title: Attentional Capture by Emotional Information in Alzheimer's Disease : an fMRI Study
Brief Title: Emotion and Attention in Alzheimer's Disease (ATEMMA)
Acronym: ATEMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2018/113; 2018-A02945-50 (Other: ID RCB)
Record Dates: First submitted 2019-05-27; First posted 2019-06-03 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer Disease
Keywords: attention; emotion; eye movements; amygdala
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young adults (Active Comparator): Participants aged between 18 and 40 years old.
  Interventions: Behavioral: Facial expression recognition task
- Healthy old adults (Active Comparator): Participants aged between 65 and 95 years old.
  Interventions: Behavioral: Facial expression recognition task
- Patients with Alzheimer's Disease (Experimental): Participants aged between 65 and 95 years old with a diagnosis of Alzheimer's Disease.
  Interventions: Behavioral: Facial expression recognition task

INTERVENTIONS:
Behavioral: Facial expression recognition task — We will present emotional expressions to participants. Their task will be to determine which emotion is expressed by each face. Participants' eye movements and brain activity will be recorded while they explore the face.

SUMMARY:
The main purpose of this study is to investigate the existence of emotional attention impairments in Alzheimer's Disease, in correlation with amygdala and attention networks alterations. To this end, functional and structural neuroimaging will be used. A face expression recognition task, along with eyetracking, will be used to assess emotional attention impairments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers :

  * Affiliation to social security
  * Medical examination before study participation
  * No contraindication to MRI
  * Informed consent signed
  * Young adults older than 18 years and younger than 40 years
  * Healthy old adults older than 65 years and younger than 95 years
  * Visual acuity allowing normal perception of stimuli or corrected to normal vision
* Patients with Alzheimer's Disease :

  * Affiliation to social security
  * Medical examination before study participation
  * No contraindication to MRI
  * Informed consent signed
  * Patients with Alzheimer's Disease at mild or moderate stage (National Institute on Aging and Alzheimer's Association criteria), diagnosed at Grenoble CMRR (Centre Mémoire de Ressources et de Recherche)
  * Patients older than 65 years and younger than 95 years
  * MMSE (Mini-Mental State Examination) > 18/30
  * Ability to understand study instructions and give an informed consent
  * Visual acuity allowing normal perception of stimuli or corrected to normal vision

Exclusion Criteria:

* Every participant having a vascular stent implanted less than 6 weeks before study
* Every participant having a biomedical material implanted that is considered "unsafe" in the list: http://www.mrisafety.com/TheList_search.asp
* Every acquisition procedure not respecting required conditions by the "conditional" usage in a participant having a biomedical material implanted that is considered "conditional" in the list: http://www.mrisafety.com/TheList_search.asp
* Every subject having a biomedical material such as a cardiac, neuronal or sensorial stimulator (cochlear implant because of demagnetization, electrode heating or artefact risk) or a ventricular drain without trained medical or paramedical support during MRI for these participants
* Ferromagnetic object inside the eye or the skull, close to nervous structures (displacement and complications risk such as eye or brain damage)
* Claustrophobia
* Psychiatric (e.g., bipolar disorder) or neurological pathology (e.g., epilepsy, Parkinson's Disease) other than Alzheimer's Disease
* Non cooperating participant
* Severe and uncontrolled affection: cardiac, respiratory, haematological, renal, hepatic, cancerous
* Participation to other research protocols with exclusion period or MRI during the past weel
* Drug therapy likely to modulate brain activity : neuroleptics, lithium, etc...
* Alcohol ingestion before study
* Participants concerned by articles L1125-5 to L1121-8 of CSP (Code de la Santé Publique) (pregnant or nursing women, underage or protected adult, person under administrative or judicial oversight
* Participant receiving more than 4500 euros for his participation to other studies involving human person during the past 12 months before this study
* Participant unable to be contacted in case of emergency
* Inability to understand study instructions or give an informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Classic recognition score | 1 hour
  Facial expression recognition score (%)
Classic fixation time faces | 1 hour
  Fixation time on eyes as measured with eyetracking (ms)
Fixation time scenes | 30 mn
  Fixation time on emotional scenes outside of MRI
Classic fMRI activity | 2 hours
  fMRI activity in amygdala and emotional attention networks during face exploration and resting-state

SECONDARY OUTCOMES:
Alternative recognition score | 1 hour
  Facial expression recognition score (%) during an alternative task designed to encourage focus on the eyes
Alternative fixation time faces | 1 hour
  Fixation time on eyes as measured with eyetracking (ms) during this alternative task.
Alternative fMRI activity | 2 hours
  fMRI activity in amygdala and emotional attention networks during this alternative task

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, La Tronche, France

IPD SHARING:
Plan to Share IPD: No